CLINICAL TRIAL: NCT01517906
Title: Developing Identity: An Eating Disorder Nursing Therapy
Brief Title: Developing Identity: An Eating Disorder Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Karen Farchaus Stein, Professor of Nursing, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01NR005277 (NIH)
Record Dates: First submitted 2012-01-18; First posted 2012-01-25 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Anorexia Nervosa; Bulimia Nervosa
Keywords: eating disorder behaviors; well being; functional health
MeSH Terms: conditions — Anorexia Nervosa; Bulimia Nervosa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioral counseling (Experimental)
  Interventions: Behavioral: Identity Intervention Program
- Supportive therapy (Active Comparator)
  Interventions: Behavioral: Supportive Psychotherapy for the Eating Disorders

INTERVENTIONS:
Behavioral: Identity Intervention Program — Cognitive behavioral strategies will be used by trained nurse-therapists to facilitate the participant's: a) identification of a small collection of personally meaningful and feasible desired possible selves, b) prioritization of the desired possible selves as short and long-term goals, c) identification, elaboration, implementation and evaluation of cognitive and behavioral strategies to achieve the desired possible self selected as the goal, and d) identification of internal and external barriers that interfere with achieving the possible self goal and utilization of active problem solving strategies to overcome the barriers.
  Arms: Cognitive behavioral counseling
Behavioral: Supportive Psychotherapy for the Eating Disorders — SPI is a 20-week program with a one-hour individual psychotherapy session scheduled each week. The SPI is organized in three stages: 1) Stage 1 (Sessions 1-8) including assessment of the current and past ED history, collection of personal and family history, and identification of problems contributing to the ED; 2) Stage 2 (Sessions 9-16) aims include exploration of underlying emotional problems, increased self-disclosure and expression of feelings, and fostering independence; and 3) Stage 3 (Sessions 17-20) includes continued exploration of underlying problems and implications for future behaviors and termination.
  Other Names: SPI
  Arms: Supportive therapy

SUMMARY:
The purpose of this research study is to test a new type of counseling developed to decrease symptoms of anorexia nervosa and bulimia nervosa and improve health and well-being in women with these eating disorders. At this time, the most effective form of treatment for anorexia nervosa and bulimia nervosa is cognitive behavioral therapy. However, this form of treatment leads to a complete absence of symptoms in only about 50% of persons completing the treatment program. In this study we will test the effectiveness of a new form of counseling that focuses on identifying and building personal strengths and positive views of the self as the means to decrease eating disorder symptoms and improve health. This study will involve 150 women between the ages of 18 and 35 years who currently have symptoms of anorexia nervosa or bulimia nervosa. To participate in this study, women must also be: 1) not pregnant, 2) without any other diagnosable mental disorder, 3) not currently taking medications for their eating disorder or other mental disorder symptoms, 4) not ill enough to require inpatient treatment for their eating disorder and 5) willing to refrain from seeking other treatment for their eating disorder for the duration of this study. Each participant will participate in a 20-week treatment program that includes nutritional counseling and medical care. Both of these forms of treatment are considered by the American Psychiatric Association to be essential parts of treatment for eating disorders and have been found help to reduce symptoms. In addition, participants will receive one of two types of counseling:

1. Experimental counseling that focuses on building strengths and positive self-views
2. Standard counseling that helps the participant identify and solve problems that are believed to contribute to their eating disorder symptoms.

The type of counseling that a participant receives will be determined randomly. To determine whether the experimental counseling is effective, eating disorder symptoms, psychological and functional health will be measured before the treatment begins and three times after the treatment ends (immediately after treatment ends, 6 and 12 months later). The findings of this research study are expected to contribute to the development of effective interventions to decrease eating disorder symptoms, and increase health and well-being in women with anorexia nervosa and bulimia nervosa.

ELIGIBILITY:
Inclusion Criteria:

* Anorexia nervosa
* Subthreshold anorexia nervosa
* Bulimia nervosa
* Subthreshold Bulimia nervosa
* Nonpregnant
* No prescribed psychotropic medication
* No concurrent psychiatric treatment
* No indications for inpatient treatment including suicide risk, significant metabolic or cardiac complications
* Willingness to refrain from seeking other forms of ED treatment until completing the intervention and post-treatment data collection protocols
* Negative lifetime history for schizophrenia, other DSM-IV Axis I psychotic disorders and mental retardation

Exclusion Criteria:

* Acute and chronic medical conditions other than those related to the ED
* Any other concurrent DSM-IV Axis I disorder at threshold level

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2002-04; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Interview | change from baseline to one month post-intervention
  A computerized menu-driven interview will be used to prospectively measure ED behaviors (event-triggered EMA methodology). Behaviors measured as outcomes include binge eating, purging, fasting & restricting and excessive exercise
Eating Disorder Inventory | Change from baseline to one month post-intervention
  A self-report measure of the ED attitudes associated with AN and BN that is widely used as an outcome measure in intervention studies. The inventory consists of 64 items that are used to generate eight subscale scores. In this study, the drive for thinness, body dissatisfaction and bulimia subscale scores will be used
Eating Disorder Interview | Change from baseline to 6 mos post-intervention
  A computerized menu-driven interview will be used to prospectively measure ED behaviors (event-triggered EMA methodology). Behaviors measured same as above
Eating Disorder Interview | Change from baseline to 12 months post-intervention
  A computerized menu-driven interview will be used to prospectively measure ED behaviors (event-triggered EMA methodology).
Eating Disorder Inventory | Change from baseline to 6 mos post-intervention
  A self-report measure of the ED attitudes associated with AN and BN that is widely used as an outcome measure in intervention studies. The inventory consists of 64 items that are used to generate eight subscale scores. In this study, the drive for thinness, body dissatisfaction and bulimia subscale scores will be used
Eating Disorder Inventory | Change from baseline to 12 mos post-intervention
  A self-report measure of the ED attitudes associated with AN and BN that is widely used as an outcome measure in intervention studies. The inventory consists of 64 items that are used to generate eight subscale scores. In this study, the drive for thinness, body dissatisfaction and bulimia subscale scores will be used

SECONDARY OUTCOMES:
Psychological Well-Being Scale | Baseline, immediate, 6, 12 m post-intervention
  The questionnaire measures 6 theoretically derived dimensions of psychological well-being including: Self-Acceptance, Positive Relations with Others, Autonomy, Environmental Mastery, Purpose in Life and Personal Growth. Each dimension is measured with a 14-item subscale.
SF-36 Survey | Baseline, immediate, 6 and 12 m post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Karen F Stein, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Michigan Medical Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Stein KF, Wing J, Lewis A, Raghunathan T. An eating disorder randomized clinical trial and attrition: profiles and determinants of dropout. Int J Eat Disord. 2011 May;44(4):356-68. doi: 10.1002/eat.20800. PMID 21472754
- [Derived] Stein KF, Corte C, Chen DG, Nuliyalu U, Wing J. A randomized clinical trial of an identity intervention programme for women with eating disorders. Eur Eat Disord Rev. 2013 Mar;21(2):130-42. doi: 10.1002/erv.2195. Epub 2012 Sep 27. PMID 23015537